CLINICAL TRIAL: NCT01465737
Title: Importance of Cohort and Histologic Type for Secular Trends in Rising Incidence and Different Survival of Uterine Cancer -a Taiwan Population-based Registry From 1979 to 2008
Brief Title: Epidemiology of Uterine Cancer in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201103107RC
Record Dates: First submitted 2011-10-26; First posted 2011-11-07 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Uterine Cancers
Keywords: epidemiology; uterine cancer; Taiwan
MeSH Terms: conditions — Uterine Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with uterine cancer: All patients diagnosed with uterine cancer in Taiwan between 1979-2008
  Interventions: Other: Histologic types

INTERVENTIONS:
Other: Histologic types — evaluate survival among different histologic types

SUMMARY:
Endometrial cancer is the second most common gynecologic cancer in Taiwan. Two types of endometrial cancer may be distinguished by standard clinicopathologic criteria; type I tumors are of low grade, endometrioid histology, estrogen related, and have a good prognosis, whereas type II tumors are high grade, of non-endometrioid histologies, unrelated to estrogen, and have a poor prognosis. Several clinicopathological parameters were reported to correlate with prognosis of endometrial cancer including tumor FIGO stage, cell type, cytological grading, depth of myometrial invasion, tumor size, lymph node status, and etc. However, there is no epidemiologic data of endometrial cancer in Taiwan. So the investigators propose this study to use Taiwan registry database provided by Department of Health to analyze the epidemiology and prognosis of uterine cancer patients in Taiwan.

DETAILED DESCRIPTION:
Study population To evaluate the epidemiology and prognosis of uterine cancer in Taiwan, we will conduct a nationwide analysis through linking national cancer registry database. Every citizen in Taiwan has a life-long identification number to link individual information, including health status. The Taiwan household registry database provided by Department of Health will be the source population. National household registry and death certificate will be adopted to ascertain the live status of study subjects, and provided individual demographic characteristics. All individual linkages between databases will be conducted according to the study protocols, i.e. databases will be linked by corresponding identification number, name (Chinese characters) and birthday, and all data included in this study will be analyzed without individual identification information. The agreement of utilizing the databases in the study was obtained from the Bureau of Health Promotion in Taiwan.

Incident and death cases ascertainment Patients with uterine cancer, including uterine carcinoma, uterine sarcoma … etc., will be identified from computerized linkage to the Taiwan national cancer registry with International Classification of Diseases for Oncology Third Edition T-code C540-C543. Histological types will be identified from morphology code in the cancer registry database. Women affected by uterine cancer and found death due to uterine cancer (International Classification of Diseases 9th edition code 182) in deaths certificate will be defined as death cases.

Statistical Analyses The numbers of person-years at risk of developing and dying for uterine cancer will be calculated. Incidence rates will be calculated by dividing the number of uterine cancer cases by the person-years at risk of developing uterine cancer. Mortality rates will be calculated by dividing the number of uterine cancer deaths by the person-years at risk of dying from uterine cancer. The association between mortality and age, histology, time periods will be estimated through Kaplan-Meier survival analysis and Cox's proportional hazards model. It is defined as significant difference statistically when p value is less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* All uterine cancer patients in Taiwan between 1979-2008

Exclusion Criteria:

* nil

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All uterine cancer patients in Taiwan between 1979-2008
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From diagnosis of uterine cancer to death or last date of linked data available from the Taiwan Cancer Registry or Death Certification Profile
  The follow-up of each participant (in personyears) was calculated from the date of enrollment to the date of uterine cancer diagnosis, date of death, or last date of linked data available from the Taiwan Cancer Registry or Death Certification Profile, whichever came first until December 31, 2010.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Fang Cheng, Professor, Principal Investigator — Department of Obstetrics and Gynecology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan